CLINICAL TRIAL: NCT05116267
Title: A Retrospective, Multicenter Study to Assess Effectiveness and Safety Outcome in Patients With Non-valvular Atrial Fibrillation (NVAF) Treated by Apixaban Using Harmonized and Federated Hospital Electronic Health Records (EHRs) in Belgium (PROVECT Study).
Brief Title: Assessment of the Effectiveness and Safety Outcome in Patients With Atrial Fibrillation Treated by Apixaban in Belgium
Acronym: PROVECT
Status: Withdrawn | Type: Observational
Why Stopped: Protocol is not feasible based on the available hospital records
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B0661166; PROVECT Study (Other: Alias Study Number)
Record Dates: First submitted 2021-09-22; First posted 2021-11-10 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Atrial Fibrillation
Keywords: Non-valvular atrial fibrillation; Belgium; Apixaban; NVAF
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
The PROVECT study is a retrospective, multicentre study assessing the effectiveness and the safety outcomes in patients with non-valvular atrial fibrillation (NVAF) treated by apixaban between 2015 and 2019 (5 years follow up). The study will use harmonized and federated hospital electronic health records (EHRs) from 10 Belgian hospitals. Outcomes of interest are major bleeding events leading to hospitalization (safety), stroke and systemic thromboembolic events (effectiveness), and all-cause mortality (as an exploratory endpoint, and after confirming the data availability because the death events are not always recorded into hospital EHRs). The study will analyse the outcomes by patient characteristics including the age groups focusing on elderly, thromboembolism risk factors (CHAR2RDSR2R-VASc score), bleeding risk factors (HAS-BLED score), comorbidities (Deyo-Charlson Comorbidity Index, DCCI) score and frailty.

DETAILED DESCRIPTION:
Apixaban is an antithrombotic agent that directly inhibits factor Xa, and which has obtained market authorization in the indication "prevention of stroke and systemic embolism in patients with non-valvular atrial fibrillation (AF), with one or more risk factors, such as prior stroke or transient ischaemic attack (TIA), age ≥75 years, hypertension, diabetes mellitus, and symptomatic heart failure (NYHA ≥ class II)." Among other direct oral anti-coagulants (DOACs) only apixaban has shown a triple beneficial profile (on stroke/systemic embolisms, major bleedings, and all-cause mortality) supported by data from pivotal randomized clinical trials (RCTs). This differentiation has been consistently found in multiple real-world data (RWD) studies including the NAXOS study in France5 and the ARISTOPHANES study in US particularly in terms of incidence of major bleedings for apixaban vs. others DOACs or vitamin K antagonists (VKAs). Although such data can be generalized to different populations, healthcare professionals in Belgium and healthcare authorities have been frequently requesting local scientific data to support the effectiveness and safety outcomes in patients treated by apixaban in local Belgium settings. This scientific data gap is particularly evident for routine care data allowing to understand the apixaban use patterns in the Belgian poly-medicated, frail and new patients starting an apixaban treatment. The PROVECT study aims to address this particular local data gap and its results may help to guide practical clinical decisions .

ELIGIBILITY:
Inclusion Criteria:

* is 18 years or older at the index date.
* had ≥1 apixaban prescription during the study period from January 1st, 2015 to December 31, 2019.
* had ≥1 medical diagnosis for Atrial Fibrillation, AF (International Classification of Diseases, 10th Revision, Clinical Modification [ICD-10-CM]10 diagnosis codes I48.0, I48.1X, I48.11, I48.19, I48.2X, I48.20, I48.21, I48.9X, I48.91, I49.1) any time before or on index date
* had >1 encounter (visits, prescriptions, etc) within the EHRs.

Exclusion Criteria:

* Medical EHRs indicating a diagnosis code indicative of rheumatic mitral valvular heart disease, mitral valve stenosis (ICD-10-CM diagnosis codes I05.x, I06.x, I07.x, I08.x, I34.x, I35.x, I36.x, I37.x, I38.x, I39.x, I37.x, Q23.x) during the 12-month baseline period,
* Medical EHRs indicating a diagnosis code of VTE (DVT: ICD-10-CM codes: I80.xx, I81.xx, I82.xx, I82.40x, I82.41x, I82.42x, I82.43x, I82.44x, I82.49x, I82.4Yx, I82.4Zx, I82.5xx, I82.51x, I82.52x, I82.53x, I82.54x, I82.55x, I82.56x, I82.59x, I82.5Yx, I82.5Zx, I82.62x, I82.72x, O22.0x, O22.2x, O22.3x; or PE: ICD-10-CM codes I26.01, I26.02, I26.09, I26.90, I26.92, I26.93, I26.94, I26.99) during the 12-month baseline period,
* Medical EHRs indicating a diagnosis (ICD-10-CM) or procedure code (International Classification of Diseases, 10th Revision, Procedure Coding System [ICD-10-PCS]10) of transient AF, or cardiac surgery: Heart valve replacement/transplant: 02YA0Zxx, 02RF0xx, 02RJ0xx, 02RG0xx, 02RH0xx, Z95.2, Z95.3, Z95.4; Pericarditis: I00, I01, I02, I24.1, I30.x, I31.x, I32*coding first the associated cause/etiology; Hyperthyroidism and Thyrotoxicity: E05.0, E05.1, E05.2, E05.3, E05.4, E05.8, E05.9) during the 12-month baseline period;
* Medical EHRs indicating pregnancy during the study period (ICD-10-CM diagnosis codes O00-O9A, Z31, Z32, Z33, Z34, Z36, Z37, Z38, O20-O29, ICD-10 CPS code 109xxx, 10Axxx, 10Dxxx, 10Exxx, 10Hxxx, 10Pxxx, 10Sxxx);
* Medical EHRs indicating diagnosis or procedure for hip/knee replacement surgery within 6 weeks prior to index date (0SR90xx, 0SRA0xx, 0SRB0xx, 0SRC0xx, 0SRD0xx, 0SRE0xx, 0SQ0xx, 0SQB0xx, 0SQB0xx, 0SQB0xx)
* Patients with a prescription for >1 anticoagulants at index date.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study is an observational retrospective cohort generated from the Belgian hospitals EHRs. The cohort will consist in anticoagulant (AC)-naive patients (patients that did not receive other oral AC 6 months prior to the apixaban treatment initiation) and AC-experienced patients (patients treated by AC before the inclusion date) diagnosed with non-valvular AF.
  The study will cover the period from 01/01/2015 to 31/12/2019 (i.e. maximum of 5 years follow up, noting that all patients will not have this follow up).
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Event Rate of Stroke/Systemic Embolism Requiring Hospitalization: Apixaban treated patients | Up to 60 months
  StroStroke/SE will be identified using hospital EHR which had a stroke/SE diagnosis code as the first listed ICD-10-CM diagnosis code. (Codes list defined) Stroke/SE will be classified into 3 categories: ischemic stroke, hemorrhage stroke, and SE. Time to stroke will be defined as the number of days from the index date to the occurrence of the first stroke/SE requiring hospitalization
Event Rate of Major Bleeding Requiring Hospitalization: Apixaban treated patients | Up to 60 months
  Major bleeding will be identified using hospital EHR which had a bleeding diagnosis code as the first listed ICD-10-CM diagnosis or procedure code (Code list defined). Time to major bleeding will be defined as the number of days from the index date to the occurrence of the first major bleeding event requiring hospitalization
Event Rate of Gastrointestinal (GI) Bleeding Requiring Hospitalization: Apixaban treated patients | Up to 60 months
  Event rate was defined as number of events divided by 100 participant-years for first occurrence of GI bleeding events after index date was reported. GI bleeding requiring hospitalization was identified using hospital claims which had a GI bleeding ICD code (Code list defined). Index date = the first prescription date of study drugs during intake duration.
Event Rate of Intracranial Hemorrhage Requiring Hospitalization: Apixaban treated patients | Up to 60 months
  Event rate was defined as number of events divided by 100 participant-years for first occurrence of intracranial hemorrhage events after index date was reported. Intracranial hemorrhage requiring hospitalization was identified using hospital claims which had an intracranial haemorrhage ICD code (Code list defined) and brain CT or MRI codes. Index date = the first prescription date of study drugs during intake duration
Event Rate of Other Bleeding Requiring Hospitalization: Apixaban treated patients | Up to 60 months
  Event rate was defined as number of events divided by 100 participant-years for first occurrence of other bleeding events after index date was reported. Other bleeding requiring hospitalization was identified using hospital claims which had other bleeding ICD code (Code list defined). Index date = the first prescription date of study drugs during intake duration.
Mortality rates | Up to 60 months
  Patients who died during a hospitalization during the follow-up period will be labelled by binary indicators.

SECONDARY OUTCOMES:
Rate of discontinuation | Up to 60 months
  Discontinuation is defined as the first day of a period of at least 30 consecutive days (grace period) in which 0 days' supply for the index OAC is detected. Sensitivity analysis with 60-day grace period will be included. The date of discontinuation will be the end date of the last filled prescription before the treatment gap. The mean and median (days) duration of treatment before discontinuation will be calculated.
Time-to-discontinuation | Up to 60 months
  Time to discontinuation will be defined as the number of days from the date of index apixaban prescription to the date of discontinuation.
Hospital Length of Stay (LOS) | Up to 60 months
  Length of stay will be defined as the number of days a patient received care during an inpatient stay. LOS will be a continuous and categorical variable.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Site, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B0661166